CLINICAL TRIAL: NCT00261040
Title: Minimally Invasive Surgery of the Hip: A Randomized Study
Brief Title: Minimally Invasive Surgery of the Hip Versus Standard Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OHREB 2003211-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Hip Arthroplasty; Osteoarthritis
Keywords: Osteoarthritis; Total Hip Arthroplasty; Minimally Invasive Surgery
MeSH Terms: conditions — Osteoarthritis | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Surgery (MIS) (Active Comparator): In minimally invasive surgery, the surgeon makes a shorter incision (about 10 cm or less) along the side of the thigh and replaces the hip through this smaller incision. The surgeon is able to do the surgery through a shorter incision by using special instruments which can guide him or her.
  Interventions: Procedure: Minimally Invasive Surgery
- Standard Surgery (Sham Comparator): The standard way an orthopaedic surgeon performs a hip replacement surgery is that they make a long incision (about 20 cm) down the side of the thigh and then replaces the hip joint through this long incision
  Interventions: Procedure: Standard Surgery

INTERVENTIONS:
Procedure: Minimally Invasive Surgery — In minimally invasive surgery, the surgeon makes a shorter incision (about 10 cm or less) along the side of the thigh and replaces the hip through this smaller incision. The surgeon is able to do the surgery through a shorter incision by using special instruments which can guide him or her.
  Arms: Minimally Invasive Surgery (MIS)
Procedure: Standard Surgery — The standard way that an orthopaedic surgeon performs a hip replacement surgery is that they make a long incision (about 20 cm) down the side of the thigh and then replaces the hip joint through this long incision.
  Other Names: non applicable
  Arms: Standard Surgery

SUMMARY:
The purpose of this study is to determine if there is a difference in terms of length of hospital stay and post-operative outcomes between patients whose total hip replacement surgery is performed with a minimally invasive versus standard surgical approach.

DETAILED DESCRIPTION:
Traditional techniques for total hip arthroplasty (THA) require complete visualization of the acetabulum and proximal femur since anatomic landmarks are crucial for correct orientation of the prosthetic components. All surgeons are taught that a wide surgical exposure is one of the most important factors in performing successful THA. Traditionally, it was impossible to achieve accurate fixation and orientation of the components without complete visualization of bony landmarks. These extensile exposures facilitate accurate implant alignment, but at the expense of more extensive soft tissue dissection. Little clinical research has been undertaken to relate the surgical approach to postoperative complications or patient function. Furthermore, despite the good overall results of THA, the recovery time to improved function can be lengthy. Blood loss is expected to be directly related to the extent of the surgical exposure and to influence patients outcomes. Based upon these facts, an important principle of arthroplasty surgery is to minimize the amount of soft tissue trauma while being able to achieve the surgical goal of reconstructing the arthritic hip joint. By definition, minimally invasive surgical (MIS) procedures result in less soft tissue disruption, which in turn should reduce pain, expedite healing, decrease recovery time, and potentially reduce the number of associated complications.

ELIGIBILITY:
Inclusion Criteria:

BMI > 30 kg/m2 No prior ipsilateral hip surgery Osteoarthritis

Exclusion Criteria:

Patients with grossly distorted bony anatomy whereby standard implants are contraindicated; i.e. congenital dysplasia of the hip, proximal femoral abnormalities, etc

Rheumatoid Arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kim, MD, Principal Investigator — OHRI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient recruitment occurred at the Ottawa Hospital (General Campus) by one of two co-investigator surgeons trained in MIS of the hip. Randomization occurred on the day of surgery in order to minimize the potential number of dropouts.
Period: Overall Study
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcomes
Description: Hospital length of stay
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Number analyzed (Participants) | 18 | 19
Days | 5.39 (1.819) | 5.74 (1.522)

2. Secondary Outcome: Harris Hip Score
Description: Questionnaire to measure health outcome status. An index score of 100 is the highest score and is indicative of better outcome, while 0 is the lowest score and indicative of worse outcome. With regards to health, a score between 90-100 is considered "Excellent." 80-89 is considered "Good." 70-79 is considered "Fair." Less than 70 is considered "Poor."
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Number analyzed (Participants) | 20 | 20
units on a scale | 90.4031 (8.92579) | 90.3011 (12.54267)

3. Secondary Outcome: Change in Timed Get-up-and-Go Test (TUG)
Description: A timed assessment to assess a participants mobility. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. A faster time is indicative of better mobility, while a slower time is indicative of worse mobility.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Number analyzed (Participants) | 20 | 20
seconds | 11.01 (4.937) | 12.03 (2.639)

4. Secondary Outcome: Operating Time Duration
Description: Duration of the surgical procedure
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Number analyzed (Participants) | 20 | 20
minutes | 95.20 (22.94) | 87.70 (23.63)

5. Secondary Outcome: Estimated Blood Loss
Description: Estimated blood loss during the operative procedure
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: Millilitres (mL)
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Number analyzed (Participants) | 20 | 20
Millilitres (mL) | 460 (215.578) | 462.50 (152.069)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Minimally Invasive Surgery (MIS) | Standard Surgery
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minimally Invasive Surgery (MIS) (N=20) | Standard Surgery (N=20)
Patient mortality (Cardiac disorders) | 1 | 0 — Patient experienced an unrelated acute coronary syndrome and passed away in hospital.
Myocardial Infarction (Cardiac disorders) | 1 | 0 — Patient experienced a myocardial infarction post-surgery, but recovered.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minimally Invasive Surgery (MIS) (N=20) | Standard Surgery (N=20)
Operative Complication (Nervous system disorders) | 0 | 1 — Femoral nerve palsy - a known possible complication of total hip replacement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No